CLINICAL TRIAL: NCT02524847
Title: Single-Arm Study to Assess the Efficacy of UVADEX® (Methoxsalen) Sterile Solution in Conjunction With the THERAKOS® CELLEX® Photopheresis System in Pediatric Patients With Steroid-Refractory Acute Graft-vs-Host Disease (aGvHD)
Brief Title: Methoxsalen and Extracorporeal Photopheresis (ECP) for the Treatment of Pediatric Participants With Steroid Refractory Acute Graft Versus Host Disease
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Therakos, Inc., a Mallinckrodt Company (Industry)
Responsible Party: Sponsor
Organization: Mallinckrodt (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TKS-2014-001
Record Dates: First submitted 2015-08-13; First posted 2015-08-17 (Estimated); Results first posted 2020-09-11 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-07

CONDITIONS: Steroid Refractory Acute Graft Versus Host Disease
MeSH Terms: interventions — Methoxsalen; Photopheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Methoxsalen with ECP (Experimental): Participants receive methoxsalen 20 µg/ml in conjunction with ECP procedure three times per week for Weeks 1 to 4, and two times per week for Weeks 5 to 12.
  Interventions: Drug: Methoxsalen; Procedure: Extracorporeal Photopheresis (ECP)

INTERVENTIONS:
Drug: Methoxsalen — Sterile solution used in conjunction with photopheresis procedure.
  Other Names: UVADEX®
Procedure: Extracorporeal Photopheresis (ECP)
  Other Names: THERAKOS® CELLEX® Photopheresis System

SUMMARY:
This is a single-arm, open-label, multicenter study of the efficacy of UVADEX® (methoxsalen) Sterile Solution in conjunction with THERAKOS® CELLEX® Photopheresis Systems (ECP) in pediatric participants with steroid-refractory aGvHD. The study is composed of Screening, Treatment, and Follow-up Periods.

DETAILED DESCRIPTION:
Screening:

After the informed consent/assent form (ICF) is signed, the screening assessments will be performed in a single visit to establish the eligibility of the participant, based on inclusion and exclusion criteria, as well as aGvHD grading. Scheduling of the first week of ECP treatments and the arrangements for availability of typed and cross-matched donor packed red blood cells (PRBCs) for transfusion, if required, will be made in advance of participants entering the Treatment Period.

Treatment Period:

Once eligibility is established, participants will enter the 12-week ECP Treatment Period. The availability of typed and cross-matched donor PRBCs for transfusion during treatment, if needed, should be established prior to the scheduling of ECP treatments.

Participants will be allowed to continue standard aGvHD prophylaxis regimens (e.g., cyclosporine, tacrolimus, methotrexate, mycophenolate mofetil) without the addition of new therapies. Participants will be allowed to discontinue prophylaxis regimens for reasons of toxicity, and will also be allowed to switch to another prophylaxis medication within the same class (e.g., the calcineurin inhibitors cyclosporine and tacrolimus) for reasons of toxicity.

All participants enrolled in this trial will have received corticosteroids for the treatment of aGvHD. After entering the treatment period on study, tapering of steroids by total weekly decrements of 12.5% to 25% of the steroid dose at initiation of ECP therapy is permitted after a sustained response of aGvHD has been observed for at least 3 consecutive days, with the suggested goal to decrease the starting steroid dose by at least 50% 4 weeks after initiation of ECP.

Follow-Up Period:

After completion of the 12-week Treatment Period, participants may continue ECP treatment on commercial product at the Principal Investigator's discretion. Acute GvHD status will be assessed 4 weeks after completion of the Treatment Period. Participant survival will be assessed by passive follow-up (chart review) 26 weeks after initiation of ECP treatment.

ELIGIBILITY:
Inclusion:

1. Male or female 1 to 21 years of age at the time of consent
2. Steroid-refractory grade B-D aGvHD.

   * Steroid-refractory is defined as a failure to respond to steroid treatment, with failure to respond defined as any grade B-D (IBMTR grading) aGvHD that shows progression ≥ 3 days, or no improvement by 5 days of treatment with 2 mg/kg/day methylprednisolone or equivalent in participants with lower gastrointestinal (GI) or liver disease, or skin disease associated with bullae. Grade D organ involvement will be limited to skin and liver.
   * Steroid refractory may also be defined as a failure to respond to 1 mg/kg/day of methylprednisolone or equivalent in participants with disease confined to upper GI disease or lesser degrees of skin GvHD
   * Participants with lack of complete response after 2 weeks of steroid treatment
3. A Lansky scale Performance Status score ≥ 30
4. Laboratory values are within the following limits, assessed within 3 days of the first study treatment:

   * Absolute neutrophil count > 0.5 × 10^9/liter (L)
   * Creatinine level < 2 times the upper limit of normal
5. For participants with isolated upper GI symptoms, pre-Screening biopsy results to confirm diagnosis of aGvHD
6. Female participants of childbearing potential and nonsterilized males who are sexually active with a female partner must be practicing highly effective, reliable, and medically approved contraceptive regimen throughout their participation in the study and for 3 months following the last ECP treatment. Or, for the US only, abstinence may be used in place of an approved contraceptive regimen. Females of childbearing potential are those who have reached the onset of menarche, or 8 years of age, whichever comes first. Approved contraceptive methods for female participants of childbearing potential or nonsterilized males who are sexually active with a female partner are as follows:

   * Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository
   * Established use of oral, injectable, or implanted hormonal methods of contraception.
   * Placement of an intrauterine device or intrauterine system
7. Signed informed consent/assent is obtained before conducting any study procedures; the parent, legal guardian, or legally authorized representative of a minor must also provide written informed consent

Exclusion:

1. Currently enrolled in another clinical trial for the treatment of aGvHD
2. Use of any experimental regimens or medication(s) for aGvHD treatment
3. Treatment with > 2.0 mg/kg/day of methylprednisolone equivalents for aGvHD within 30 days prior to the first study treatment
4. Overt signs of relapse of the underlying condition
5. Uncontrolled viral, fungal, or bacterial infection
6. Platelet count < 20.0 × 10^9/L, despite platelet transfusion
7. Inability to tolerate the extracorporeal volume shifts associated with ECP treatment
8. Uncontrolled GI bleeding
9. Veno-occlusive liver disease
10. Life expectancy < 4 weeks
11. Participant requires invasive ventilation or vasopressor support
12. Known human immunodeficiency virus (HIV) or hepatitis B or C virus infection (proof of seronegativity within 6 months of screening is required)
13. Known allergy or hypersensitivity to methoxsalen, Uvadex, or its excipients
14. Known hypersensitivity and allergy to heparin and Anticoagulant Citrate Dextrose Formula-A (ACD-A)
15. Co-existing photosensitive disease (e.g., porphyria, systemic lupus erythematosus, albinism) or aphakia
16. Coagulation disorders that cannot be corrected with simple transfusion
17. Co-existing melanoma, basal cell, or squamous cell skin carcinoma
18. Previous splenectomy
19. White blood cell count greater than 25,000 cubic millimeter (mm^3)
20. Currently being treated with any systemic immunosuppressive or biologic therapy for the treatment of a medical condition other than aGvHD
21. Female participant is breastfeeding or pregnant
22. Any medical concerns that may pose risk to the participant
23. Any psychological, familial, sociological, and/or geographical condition that may potentially hamper compliance with the study protocol and follow-up schedule

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 29 (Actual)
Dates: Start 2016-01-20 (Actual); Primary Completion 2019-07-16 (Actual); Study Completion 2019-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Team Leader, Study Director — Mallinckrodt
Locations (32):
- United States (17):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Yale University, New Haven, Connecticut
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta, Emory - Children's Center, Atlanta, Georgia
  - Lurie Children's Hospital, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - St. Louis Children's Hospital, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - University Hospitals Rainbow Babies & Children's, Cleveland, Ohio
  - Cleveland Clinic Children's, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Vanderbilt University Medical Center - Ingram Cancer Institute, Nashville, Tennessee
  - MD Anderson Cancer Care Center, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- St Anna Kinderspital, Vienna, Austria
- France (2):
  - Hopital Necker Enfants Malades, Paris
  - Hôpital universitaire Robert Debré, Paris
- Germany (4):
  - Universitätsklinikum Leipzig, Klinik und Poliklinik für Kinder- und Jugendmedizin, Abteilung für Hämatologie und Internistische Onkologie, Leipzig
  - Klinikum rechts der Isar, TU München, Klinik- und Poliklinik für Kinder- und Jugendmedizin, Kinderklinik München Schwabing, München
  - University Hospital Tuebingen, Tübingen
  - Universitaetsklinikum Ulm, Kinder- und Jugendmedizin, Ulm
- United St Istvan and St Laszlo Hospital, Budapest, Hungary
- Italy (2):
  - U.O.C. Clinica di Oncoematologia Pediatrica Azienda Ospedaliera di Padova, Padua
  - Pediatric Hospital Bambinu Gesu Rome, Rome
- Spain (4):
  - Vall d'Hebron University Hospital, Barcelona
  - Hospital Infantil Universitario "Nino Jesus", Madrid
  - University Hospital Salamanca, Salamanca
  - Hospital LA FE, Valencia
- Great North Children's Hospital (RVI), Newcastle, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Because we work in the rare disease space, to eliminate risk of patient identification we do not share individual patient data.
  We post summary aggregate results for applicable clinical trials in the registry, and statistical endpoints and discussion in publications; with each referencing the other.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were recruited by multiple treatment centers in the United States and Europe
Groups:
- Methoxsalen With ECP: Participants receive methoxsalen 20 µg/ml in conjunction with extracorporeal photopheresis (ECP) procedure three times per week for Weeks 1 to 4, and two times per week for Weeks 5 to 12.
Period: Overall Study
Arm/Group | Methoxsalen With ECP
Started | 29
Completed Treatment Up to Week 12 (Includes participants who received ECP treatments up to and including Week 12) | 14
Started Second Line Treatment | 5
Completed | 15
Not Completed | 14
Not completed — Adverse Event | 4
Not completed — Unsatisfactory Therapeutic Effect | 4
Not completed — Condition no Longer Requires Treatment | 4
Not completed — Death | 1
Not completed — Reason not Specified | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants who receive any amount of study drug.
Arm/Group | Methoxsalen With ECP
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.6 (5.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1
  Black or African American | 2
  White | 22
  Other | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving Overall Response (OR) Using the Modified International Bone Marrow Transplant Registry (IBMTR) Severity Index at Week 4
Description: OR using the modified IBMTR Severity Index is defined as complete response (CR) + partial response (PR) as follows:
  * CR: complete resolution of all signs and symptoms of aGvHD in all evaluable organs without addition of next-line systemic treatment
  * PR: improvement of 1 stage in 1 or more aGvHD target organs without progression in others and without addition of next-line systemic treatment
Time Frame: 4 weeks
Population: All participants
Measure: Count of Participants; unit: Participants
Arm/Group | Methoxsalen With ECP
Number analyzed (Participants) | 29
Participants | 16
Statistical Analysis 1: Comparison: Methoxsalen With ECP; Test type: Other; p < .001, t-test, 2 sided; 2-sided p-value for testing the null hypothesis H0: Standard therapy has a CR+PR rate = 10% after 4 weeks, using the exact Binomial test; Overall response rate (%) = 55.2, 95% CI 2-sided [35.7 to 73.6]

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Clinically significant changes in vital signs, laboratory values and investigations are reported as adverse events. Summary data are provided below, with details listed in the adverse events module.
Time Frame: 16 weeks
Population: All participants
Measure: Count of Participants; unit: Participants
Arm/Group | Methoxsalen With ECP
Number analyzed (Participants) | 29
Participants
  Any serious AE | 12
  Non-serious TEAE at 5% threshold | 17
  Death for any cause | 3

3. Secondary Outcome: Percentage of Participants Achieving Overall Response (OR) Using Modified IBMTR Severity Index at Week 8
Description: as for outcome 1
Time Frame: 8 weeks
Population: Evaluable Participants (Participants with appropriate efficacy data at the given time point)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Methoxsalen With ECP
Number analyzed (Participants) | 19
percentage of participants | 73.7 [48.8 to 90.9]

4. Secondary Outcome: Percentage of Participants Achieving Overall Response (OR) Using Modified IBMTR Severity Index at Week 12
Description: as for outcome 1
Time Frame: 12 weeks
Population: Evaluable Participants (Participants with appropriate efficacy data at the given time point)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Methoxsalen With ECP
Number analyzed (Participants) | 14
percentage of participants | 78.6 [49.2 to 95.3]

5. Secondary Outcome: Duration of Response (Days) Within 16 Weeks Using Modified IBMTR Severity Index
Description: Duration of first response is presented for patients whose disease progressed.
  Duration of response is defined in the following way:
  Patients whose response failed: Date at which 1st disease progression occurs - date of 1st response +1.
  Patients whose response did not relapse: Date of 16 week follow-up or final assessment prior to week 16 (if patient withdrew early) - date of 1st response.
Time Frame: 16 weeks
Population: Population meeting the criterion
Measure: Median (Full Range); unit: days
Arm/Group | Methoxsalen With ECP
Number analyzed (Participants) | 18
days | 13.5 [4 to 50]

6. Secondary Outcome: Overall Response Rate (ORR) According to the Modified Glucksberg Criteria
Description: ORR is defined as the percentage of patients who achieve an overall response after 4 weeks, 8 weeks, and 12 weeks of ECP treatment according to a scoring algorithm applied to calculate the grade of aGvHD using the modified Glucksberg Criteria.
Time Frame: 4 weeks, 8 weeks, and 12 weeks
Population: All participants with a score at the given time point
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Methoxsalen With ECP
Number analyzed (Participants) | 29
percentage of participants
  Week 4: number analyzed (Participants) | 24
  Week 4 | 50 [29.1 to 70.9]
  Week 8: number analyzed (Participants) | 19
  Week 8 | 63.2 [38.4 to 83.7]
  Week 12: number analyzed (Participants) | 14
  Week 12 | 78.6 [49.2 to 95.3]

7. Secondary Outcome: Cumulative Dose of Daily Steroids
Description: Steroids administered from diagnosis of aGvHD to 12 Weeks after initiation of ECP treatment
Time Frame: From diagnosis of aGvHD to 12 Weeks
Population: All participants
Measure: Median (Full Range); unit: mg
Arm/Group | Methoxsalen With ECP
Number analyzed (Participants) | 29
mg | 1917 [192 to 6895]

8. Secondary Outcome: Number of Patients With Skin Rated as Stage 0 - 4 Using the Modified Glucksberg Criteria
Description: Number of patients whose skin was rated as Stage 0 - 4 using the modified Glucksberg criteria based on the Graft versus Host Disease (GvHD) rash - Stages are defined as 0=No GvHD rash, 1=Maculopapular rash on <25% body surface area (BSA), 2=Maculopapular rash on 25-50% BSA, 3=Maculopapular rash on >50% BSA, and 4=Generalized erythroderma plus bullous formation, which are blisters bigger than 5 mm across
Time Frame: at 4, 8 and 12 weeks
Population: All participants with scores at the given time point
Measure: Count of Participants; unit: Participants
Groups:
- All Participants: Participants receive methoxsalen 20 µg/ml in conjunction with ECP procedure three times per week for Weeks 1 to 4, and two times per week for Weeks 5 to 12.
Arm/Group | All Participants
Number analyzed (Participants) | 29
Participants
  Week 4: number analyzed (Participants) | 23
  Week 4: Stage 0 | 9
  Week 4: Stage 1 | 8
  Week 4: Stage 2 | 3
  Week 4: Stage 3 | 3
  Week 4: Stage 4 | 0
  Week 8: number analyzed (Participants) | 18
  Week 8: Stage 0 | 11
  Week 8: Stage 1 | 5
  Week 8: Stage 2 | 1
  Week 8: Stage 3 | 1
  Week 8: Stage 4 | 0
  Week 12: number analyzed (Participants) | 14
  Week 12: Stage 0 | 10
  Week 12: Stage 1 | 2
  Week 12: Stage 2 | 1
  Week 12: Stage 3 | 1
  Week 12: Stage 4 | 0

9. Secondary Outcome: Number of Patients With Liver Rated as Stage 0 - 4 Using the Modified Glucksberg Criteria
Description: Number of patients whose liver was rated as Stage 0 - 4 on the modified Glucksberg criteria - Stages are based on level of bilirubin, defined as: Stage 0 = Bilirubin < 2.0 mg/dL, Stage 1 = Bilirubin 2.0-3.0 mg/dL, Stage 2 = Bilirubin 3.1-6.0 mg/dL, Stage 3 = Bilirubin 6.1-15.0 mg/dL, and Stage 4 = Bilirubin > 15.0 mg/dL
Time Frame: at 4, 8 and 12 weeks
Population: All participants with scores at the given time point
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 29
Participants
  Week 4: number analyzed (Participants) | 21
  Week 4: Stage 0 | 19
  Week 4: Stage 1 | 1
  Week 4: Stage 2 | 1
  Week 4: Stage 3 | 0
  Week 4: Stage 4 | 0
  Week 8: number analyzed (Participants) | 13
  Week 8: Stage 0 | 13
  Week 8: Stage 1 | 0
  Week 8: Stage 2 | 0
  Week 8: Stage 3 | 0
  Week 8: Stage 4 | 0
  Week 12: number analyzed (Participants) | 12
  Week 12: Stage 0 | 12
  Week 12: Stage 1 | 0
  Week 12: Stage 2 | 0
  Week 12: Stage 3 | 0
  Week 12: Stage 4 | 0

ADVERSE EVENTS:
Time Frame: Up to 16 weeks
Arm/Group | Methoxsalen With ECP
All-Cause Mortality (participants affected / at risk) | 3/29
Serious Adverse Events (participants affected / at risk) | 12/29
Other Adverse Events (participants affected / at risk) | 17/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Methoxsalen With ECP (N=29)
Aspergilloma (Infections and infestations) | 1
Bk virus infection (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Cystitis viral (Infections and infestations) | 1
Cytomegalovirus infection (Infections and infestations) | 1
Device related infection (Infections and infestations) | 1
Hepatitis E (Infections and infestations) | 1
Pyrexia (General disorders) | 2
General physical health deterioration (General disorders) | 1
Acute graft versus host disease (Immune system disorders) | 2
Acute graft versus host disease in intestine (Immune system disorders) | 1
Acute graft versus host disease in liver (Immune system disorders) | 1
Graft versus host disease (Immune system disorders) | 1
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Cystitis haemorrhagic (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Haemorrhage intracranial (Nervous system disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Methoxsalen With ECP (N=29)
Abdominal pain (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 2
Malnutrition (Metabolism and nutrition disorders) | 2
Hypertension (Vascular disorders) | 4
Hypotension (Vascular disorders) | 3
Clostridium difficile infection (Infections and infestations) | 2
Cytomegalovirus infection (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Pyrexia (General disorders) | 3
Hypogammaglobulinaemia (Immune system disorders) | 3
Immunoglobulins decreased (Investigations) | 2
Depression (Psychiatric disorders) | 2

LIMITATIONS AND CAVEATS:
This study did have a notable limitation in its single-group study design. This may limit a more robust assessment vs standard of care alone for primary endpoint of overall response and secondary endpoints steroid sparing and disease progression.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-27): https://cdn.clinicaltrials.gov/large-docs/47/NCT02524847/Prot_SAP_000.pdf